CLINICAL TRIAL: NCT01137175
Title: Laboratory Diagnosis of of Rickettsial and Rickettsia-like Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-970216
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2011-06

CONDITIONS: Rickettsioses
Keywords: Rickettsioses; Scrub Typhus; Q fever; Typhus fever; Spotted fever; Rickettsioses reported cases
MeSH Terms: conditions — Rickettsia Infections; Scrub Typhus; Q Fever; Typhus, Endemic Flea-Borne; Spotted Fever Group Rickettsiosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The low confirmed rickettsioses cases rate may indicate the presence of rickettsiosis other than scrub typhus, murine typhus, and Q fever. The clinical presentation of rickettsiosis is variable and atypical that laboratory confirmation is necessary. This project is aimed to set up the laboratory to diagnose rickettsial and rickettsial like disease, which could help in develop rapid diagnostic kits, epidemiologic surveillance and prognostic factor.

ELIGIBILITY:
Inclusion Criteria:

* Rickettsioses reported cases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients suspect to be infected by Rickettsia pathogen
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-01

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan